CLINICAL TRIAL: NCT05272124
Title: Comparison of Hip Abductors and Quadriceps Strengthening With Quadriceps Strengthening Alone in Knee Osteoarthritis
Brief Title: Effects of Hip Abductors Strengthening In Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/RCRS/REC/00940
Record Dates: First submitted 2022-02-20; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis Knees Both

STUDY DESIGN:
Intervention Model Description: Two groups are formed. Control group and Experimental group.
Who Masked: Participant
Masking Description: Study is single blinded Randomized control Trials.patients are randomly allocated into two groups through lottery method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Abductor Strengthening (Experimental): This group received quadriceps and hip abductor strengthening along with patellar mobilization and stretching exercises.
  Interventions: Other: Hip Abductor Strengthening
- Traditional Physical Therapy (Active Comparator): This group received quadriceps strengthening along with patellar mobilization and stretching exercises.
  Interventions: Other: Traditional Physical Therapy

INTERVENTIONS:
Other: Hip Abductor Strengthening — Elastic resisted training of Hip Abductors (5-10 seconds hold) 10 repetitions x 3 sets, 3 alternate days per week.
  Elastic resisted training of Quadriceps (5-7 seconds hold) 10 repetitions x 3 sets, 3 alternate days per week.
  Static Stretching of 5 seconds hold (Calf, Hamstrings, Gluteal muscles and Iliotibial band) 10 repetitions x 3 sets, 3 alternate days per week.
  Patellar Mobilization in all four directions 10 repetitions x 3 sets, 3 alternate days per week.
  Total 18 sessions were given in 06 weeks.
  Arms: Hip Abductor Strengthening
Other: Traditional Physical Therapy — Elastic resisted training of Quadriceps (5-7 seconds hold) 10 repetitions x 3 sets, 3 alternate days per week.
  Static Stretching of 5 seconds hold (Calf, Hamstrings, Gluteal muscles and Iliotibial band) 10 repetitions x 3 sets, 3 alternate days per week.
  Patellar Mobilization in all four directions 10 repetitions x 3 sets, 3 alternate days per week.
  Total 18 sessions were given in 06 weeks.
  Arms: Traditional Physical Therapy

SUMMARY:
The aim of my study is to determine the effects of hip abductors strengthening and quadriceps strengthening in comparison with quadriceps strengthening alone in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
As the quadriceps strengthening is a keystone of exercise therapy for knee osteoarthritis. Thus is the hip abductors strengthening along with quadriceps strengthening would be added to the treatment protocol of osteoarthritis it might give more positive results, decrease pain and increase the recovery rate as well as helpful to improve the functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of single or both knees
* Kellgren Lawrence scale between 2-4

Exclusion Criteria:

* Knee valgus or varus deformity
* Hip or knee joint replacement
* Tibial osteotomy
* Any other surgery of hip or knee joint

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  Changes from baseline- The Numeric Pain Rating Scale is a self-reported, or clinician administered, measurement tool consisting of a numerical point scale from 0-10 with extreme anchors of '0-no pain' to '10-extreme pain'. The scale ranges most commonly from 0-10 or 0-100, and can be administered in written or verbal form. 0 means " no pain" ands 10 or 100 means "Worst pain imaginable"
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 weeks
  Changes from baseline- The Western Ontario and McMaster Universities Osteoarthritis Index is a tested questionnaire to assess symptoms and physical functional disability in patients with Osteoarthritis of the knee and the hip. The function dimension explores the degree of difficulty in 17 activities. Its score ranges from 0-96. 0 represents the best health status and 96 the worst possible status

SECONDARY OUTCOMES:
Five Times Sit to Stand Test (FTSST) | 6 weeks
  Changes from baseline- Five time Sit-to-Stand Test was related to lower-extremity proprioception, postural sway, strength, and visual contrast sensitivity. Various methods have been used in an attempt to determine how well older adults can rise from a chair have suggested repeating the chair rise 5 times.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Khattak Physiotherapy and Rehabilitation Center, Mansehra, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No